CLINICAL TRIAL: NCT03989479
Title: The Effectiveness of T-shaped Toothbrush in Plaque Removal and Maintaining Gingival Health Among Children
Brief Title: Effectiveness of T-shaped Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T1
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Oral Hygiene
Keywords: toothbrush; plaque removal; gingival health

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Toothbrush (Active Comparator): Brushing with conventional Kid's Soft Toothbrush, Colgate (5-9-year-old)
  Interventions: Behavioral: Brushing demonstration using conventional toothbrush
- T-shaped Toothbrush (Experimental): Brushing with T-shaped toothbrush (Denson™, Malaysia)
  Interventions: Behavioral: Brushing demonstration using T shaped toothbrush

INTERVENTIONS:
Behavioral: Brushing demonstration using T shaped toothbrush — Brushing demonstration given at baseline and reinforced at 2 weeks and 1 month
  Arms: T-shaped Toothbrush
Behavioral: Brushing demonstration using conventional toothbrush — Brushing demonstration given at baseline and reinforced at 2 weeks and 1 month
  Arms: Conventional Toothbrush

SUMMARY:
This study evaluated the effectiveness of two manual toothbrushes, the T-shaped toothbrush (Denson™, Malaysia) and a conventional toothbrush (Kid's Soft Toothbrush, Colgate) in removing plaque and maintaining gingival health among 8-10-year old children.

Brushing demonstration was provided at baseline and reinforced at 2 weeks and 1 month interval.Plaque scores and gingival scores were measured at 2 weeks and 1 month and 3 months

DETAILED DESCRIPTION:
T-shaped toothbrush (Denson™, Malaysia) was introduced that is designed to efficiently clean and reduce gingival inflammation. Unlike most common conventional manual toothbrush, this new toothbrush was designed to employ a vertical motion on all tooth surfaces which simulates the natural up and down movement of the hand, suggesting that this makes the brushing process to be more controlled and stable.

One hundred and ten participants were assigned randomly to conventional toothbrush (Kid's Soft Toothbrush, Colgate) as a control group, while another half were assigned the T-shaped toothbrush (Denson™, Malaysia) as an experimental group.

Gingival status was scored using the Loe and Silness Gingival Index 25. The amount of plaque was scored using the modified Quigley and Hein Plaque Index (TQHI) 26. Both indices were recorded at 6 sites around all the teeth (mesiobuccal, midbuccal, distobuccal, mesiopalatal, midpalatal, distopalatal). All teeth were included except teeth with prosthetic crowns or cervical restorations.

One hundred children completed the study.

ELIGIBILITY:
Inclusion Criteria:

* good systemic health
* normal motor and cognitive development

Exclusion Criteria:

* acute intraoral lesion
* history of antibiotic and/ or antiseptic therapy in the past one month
* interproximal caries or restorations
* 3 or more missing teeth in one quadrant

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Plaque score | 3 months
  Plaque score measurement performed at baseline, after 2 weeks, 1 month and 3 months.
  Plaque score measurement (amount of plaque) was recorded on both the buccal and lingual sides of all teeth using the modified Quigley and Hein Plaque Index (Turesky et al., 1970) {0-no plaque present, 1- separate flecks of plaque at the cervical margin, 2- a thin, continous band of plaque at the cervical margin, 3- a band of plaque wider than 1mm but covering less than 1/3 of the surface, 4- plaque covering at least 1/3 but less than 2/3 of the surface, 5- plaque covering more than 2/3 of the surface}. Each tooth was scored in six areas: mesiofacial, midfacial, distofacial, mesiolingual, midlingual and distolingual. The minimum and maximum score per tooth was 0 and 30. The scores for each participant was summed and divided by the total number of measurements (number of teeth scored multiplied by six). Higher scores indicated worse outcome.
Gingival status | 3 months
  Gingival status measurement performed at baseline, after 2 weeks, 1 month and 3 months.
  Gingival status (gingival inflammation) was scored using the Loe and Silness (Loe & Silness, 1963) {0-absence of inflammation, 1- mild inflammation, 2- moderate inflammation, 3- severe inflammation}. Each tooth was scored in six areas: mesiofacial, midfacial, distofacial, mesiolingual, midlingual and distolingual. The minimum and maximum score per tooth was 0 and 18. The scores for each participant was calculated by adding all the individual plaque scores and dividing this sum by the total number of measurements (number of teeth scored multiplied by six). Higher scores indicated worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Shani Ann Mani, MDS, Study Chair — Faculty of Dentistry, University of Malaya

REFERENCES:
- [Derived] Mamat N, Mani SA, Danaee M. T-shaped toothbrush for plaque removal and gingival health in children: a randomized controlled trial. BMC Oral Health. 2022 Apr 7;22(1):113. doi: 10.1186/s12903-022-02137-x. PMID 35392881

DOCUMENTS (1):
  • Informed Consent Form (2014-11-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT03989479/ICF_000.pdf